CLINICAL TRIAL: NCT00622830
Title: Phase I Study of SB-480848 (Darapladib) -A Double Blind, Randomised, Placebo-controlled, Parallel-group, Repeat Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SB-480848 in Healthy Japanese Male Subjects-
Brief Title: Phase I Study of SB-480848(Darapladib) -Repeat Dose Study in Healthy Japanese Male Subjects-
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LPL110736
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Atherosclerosis
Keywords: darapladib,; SB480848,; Japanese healthy volunteers
MeSH Terms: conditions — Atherosclerosis | interventions — darapladib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB-480848 (Darapladib)

SUMMARY:
This study is being conducted to provide safety, tolerability, PK and PD data in repeat dosing that will allow further studies with darapladib in Japanese patients

ELIGIBILITY:
Inclusion criteria:

* Healthy Japanese adult males between 20 and 64 yeas of age, inclusive.
* Healthy subjects are defined as individuals who are free from clinically significant disease as determined by their medical history, physical examination, clinical laboratory examinations, vital sign, 12-lead ECG, immunology tests and urinary drug screen test.
* Bodyweight >50 kg and body mass index (BMI) between 18.5 and 25.0 at screening.
* Subjects must be capable of providing written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Baseline QTc interval <450 msec.
* Non-smoker or ex-smoker having ceased smoking for at least 6 months.
* Clinical laboratory examination (AST, ALT, ALP and GGT) at screening are within the normal range.
* The subject is able to attend all visits and complete the study.

Exclusion criteria:

* Any clinically relevant abnormality identified on the screening physical examination, vital sign measurement, 12-lead ECG recording and/or clinical laboratory examination that is deemed by the principal investigator and/or medical monitor to make the subject ineligible for inclusion because of a safety concern.
* History of regular alcohol consumption exceeding, on average, 14 drinks/week for men (1 drink = 5 ounces (150 mL) of wine or 350 mL of beer or 1.5 ounces (45 mL) of 80 proof distilled spirits) within 6 months of screening.
* Positive for urine drug at screening.
* Positive for syphilis, HIV antibody, Hepatitis B surface antigen, Hepatitis C antibody or HTLV-1 antibody at screening.
* Use of prescription or no-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* Consumption of grapefruit juice or food within 7 days prior to the first dose of study medication.
* A history of cholecystectomy or biliary tract disease including a history of liver disease with elevated liver function tests of known or unknown etiology.
* Donation of blood in excess of 400mL within 4 months or 200mL within 1 months prior to at screening.
* History of drug abuse, or current conditions of drug abuse or alcoholism.
* Participation in a clinical study or post-marketing study with an investigational or a non-investigational product or device within 4 months of preceding the first dose of study medication.
* Participation in another clinical study or post-marketing study in which the subject is or will be exposed to an investigational or a non-investigational product or device.
* History of asthma, anaphylaxis or anaphylactoid reactions, severe allergic responses.
* The subject has an allergy for any drug or idiosyncrasy. This excludes a pollen allergy without current symptoms.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Safety/tolerability of repeat oral doses of darapladib
Primary Pharmacokinetic parameters of repeat oral doses of darapladib

SECONDARY OUTCOMES:
-Secondary PK parameters
Tmax, and t1/2 of SB-480848 and AUC, Cmax, t1/2 and Tmax of the pharmacologically active metabolite SB-553253 (as data permit)
Plasma Lp-PLA2 activity, expressed in terms of percent inhibition relative to baseline
Estimation of PK/PD parameters and their associated variability, appropriate to the final models
-PK parameters of SB553253
-description of plasma concentration-Lp-PLA2 activity inhibition relationship after repeat oral doses of darapladib. all measured same timepoints as primary
-inhibition of Lp-PLA2 activity

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ibaraki, Japan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: LPL110736 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LPL110736 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LPL110736 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LPL110736 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: LPL110736 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LPL110736 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LPL110736 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register